CLINICAL TRIAL: NCT05421065
Title: Psilocybin-Assisted vs Ketamine-Assisted Psychotherapy for Alcohol Use Disorder
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peggy C Nopoulos (Other)
Responsible Party: Sponsor-Investigator, Peggy C Nopoulos, Professor of Psychiatry, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 202205036
Record Dates: First submitted 2022-06-12; First posted 2022-06-16 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Use Disorder
Keywords: psilocybin; ketamine
MeSH Terms: conditions — Alcoholism | interventions — Psilocybin; Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Psilocybin Group (Arm 1) (Experimental)
  Interventions: Drug: Psilocybin
- Ketamine Group (Arm 2) (Active Comparator)
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Psilocybin — 1 oral dose
  Arms: Psilocybin Group (Arm 1)
Drug: Ketamine — 1 oral dose
  Arms: Ketamine Group (Arm 2)

SUMMARY:
This pilot study will collect preliminary data that measures the effects of psilocybin-assisted psychotherapy vs ketamine-assisted psychotherapy on patients struggling with alcohol use.

DETAILED DESCRIPTION:
This pilot study will be a double blind, randomized, active-comparator controlled trial with two study arms. Subjects randomized to Arm 1 (n=10) will receive individual psychotherapy sessions plus a 25mg dose of psilocybin, while Arm 2 subjects (n=10) will receive individual psychotherapy sessions and a 200mg dose of ketamine. Psychotherapy sessions will involve integrative psychotherapy modalities.

At baseline, subjects will be consented, randomized into one of the two arms, complete psychiatric and medical evaluations, and will undergo an MRI scan. The first two therapy sessions (week 1 and week 2) will be used to learn about the participant's life story, engage the patient, and evoke their reasons for wanting to change their pattern of alcohol use. At week 3, participants will undergo a psilocybin-assisted therapy session or a ketamine-assisted therapy session. The last 2 psychotherapy sessions will be focused on integration of their experiences in the drug administration session and will include a second MRI scan and more assessments. Therefore, each arm receives 4 psychotherapy sessions, and the primary difference between the groups is which drug participants receive. After the psychotherapy sessions are completed at the end of week 4, subjects will be followed weekly for 4 weeks. At the last follow-up (week 8), they will undergo a third MRI scan and a final assessment. At the conclusion of the study, those randomized to the ketamine group will be offered a psilocybin-assisted therapy session, and two follow-up/integration sessions in an open-label extension. The open-label extension will also include an additional 4 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 25-65 years old
* Male
* English fluency
* Meets criteria for DSM-V moderate or severe AUD.
* Have at least 4 heavy drinking days (5 or more standard drinks in a day) in the past 30 days.
* No history of a of cerebrovascular accident, asthma, or significant alcohol withdrawal history
* No seizure disorder, coronary artery disease, heart failure, uncontrolled hypertension, insulin-dependent diabetes
* No current substance use disorder other than AUD
* Negative drug screen (other than THC) on drug administration day
* No prescription medications classified as UGT1A9 inhibitors, UGT1A10 inhibitors, aldehyde or alcohol dehydrogenase inhibitors.
* At least a high-school level of education or equivalent (e.g. GED).
* Lived at current residence for at least 3 months.
* Family member/friend for pick-up, overnight post-drug session monitoring.
* No hallucinogen or ketamine use in past 1 year
* No self-reported, personal, or familial history of specific psychotic disorders/episodes as subjects who take psilocybin may experience a worsening and/or persistent psychotic state. Therefore, these subjects are excluded due to an abundance of caution since even a family history may create a vulnerability to psychosis.
* No serious traumatic brain injury (TBI) in the past 2 years.
* No known allergies to rescue medication (diazepam)
* Weight between 110 and 330 lbs

Exclusion Criteria:

* Drug/medication assessment that yields: nonprescription medication use, nutritional supplement, or herbal supplement (except when approved by the study investigators), medically unstable, current medication use that has significant potential to interact with study drug (e.g., antidepressants, antipsychotics, psychostimulants, treatments for addictions, other dopaminergic or serotonergic agents, lithium, anticonvulsants, or benzodiazepines).
* Psychiatric assessment that yields:1) history of severe suicide attempt, 2) current suicidality 3) first degree relative with schizophrenia or schizoaffective disorder, 4) comorbid substance use including cocaine, psychostimulant, or opioid use disorder within past 12 months and/or any use within past 30 days, 5) history of co-occurring psychotic episode/diagnosis including schizophrenia, schizoaffective disorder, schizophreniform, substance-induced psychosis, delusional disorder, or psychosis not otherwise specified, 6) high risk of adverse emotional or behavioral reaction based on the medical monitor's clinical evaluation that may also yield evidence of serious current stressors, a lack of meaningful social support, antisocial behavior, and/or serious personality disorders amongst other conditions.
* Medical assessment that yields: serious ECG abnormalities (evidence of ischemia, myocardial infarction, QTc prolongation [QTc > .045]), serious abnormalities of complete blood count or chemistries, medical conditions that would preclude safe participation (significantly impaired liver function).
* MRI contraindication (pacemaker, etc.)

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Timeline Follow-Back for Alcohol to assess change | weekly, over the course of 8 weeks
  quantifies daily alcohol use

SECONDARY OUTCOMES:
T1rho | three times (before intervention, immediately after intervention, and 4 weeks-post intervention)
  Measures biological changes in the brain
Resting state fMRI | three times (before intervention, immediately after intervention, and 4 weeks-post intervention)
  Measures biological changes in the brain

OTHER OUTCOMES:
Feasibility and acceptability of the protocol | 1 year
  Measure study's rate of attrition by recording the number of participants who withdraw from the study or are discharged from the study before completion
Feasibility and acceptability of the protocol | 1 year
  Measure frequency and nature of adverse events (AEs) through recording total number of AEs and their severity on a scale of mild to moderate to severe (1-3 scale with 3 being the worst outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Peggy C Nopoulos, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davis AK, Barrett FS, May DG, Cosimano MP, Sepeda ND, Johnson MW, Finan PH, Griffiths RR. Effects of Psilocybin-Assisted Therapy on Major Depressive Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2021 May 1;78(5):481-489. doi: 10.1001/jamapsychiatry.2020.3285. PMID 33146667
- [Background] Bogenschutz MP, Forcehimes AA, Pommy JA, Wilcox CE, Barbosa PC, Strassman RJ. Psilocybin-assisted treatment for alcohol dependence: a proof-of-concept study. J Psychopharmacol. 2015 Mar;29(3):289-99. doi: 10.1177/0269881114565144. Epub 2015 Jan 13. PMID 25586396
- [Background] Johnson M, Richards W, Griffiths R. Human hallucinogen research: guidelines for safety. J Psychopharmacol. 2008 Aug;22(6):603-20. doi: 10.1177/0269881108093587. Epub 2008 Jul 1. PMID 18593734